CLINICAL TRIAL: NCT03339648
Title: Enhancing School Safety Officers' Effectiveness Through Online Professional and Job Embedded Coaching
Acronym: MiamiSROs
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: U.S. Department of Justice (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: IRB201702520; 2017-CK-BX-0019 (Other: US Dept of Justice National Institute of Justice)
Record Dates: First submitted 2017-11-01; First posted 2017-11-13 (Actual); Last update posted 2021-02-12 (Actual); Status verified 2021-02

CONDITIONS: Bullying; School Fear; Professional Role
Keywords: School Resource Officer; Trauma Informed Care; Cultural Competency; Restorative Problem Solving; Social Emotional Learning; Professional Development; School Violence
MeSH Terms: conditions — Bullying

STUDY DESIGN:
Intervention Model Description: During the measurement period, the experimental arm will receive the intervention while the control arm continues business as usual. After all data collection, the control arm will receive the intervention.
Masking Description: All participants and study staff will be aware of which schools are in each arm.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Professional Development Enhancement (Experimental): During the measurement period, this group will receive the intervention, described below:
  Content using three of UF Lastinger Center's innovations for cost-effective teaching and learning - e-Content Clinics, Coaching, and Communities of Practice. Elements of the professional development model are as follows:
  1. E-Content Clinics- Content Clinics are offered online using digital video technology.
  2. Coaching- Coaching develops strong cadres of leaders that have profound expertise and substantial success in advancing teaching and learning outcomes. This approach uses existing personnel to reinforce and deepen learning through online professional development by embedding it in day-to-day activities.
  3. Online Community of Practice- This scalable online platform allows users to create virtual communities of practice designed to strengthen the learning and collaboration network.
  Interventions: Behavioral: Professional Development Enhancement
- Control- Delayed Intervention (Active Comparator): This arm will continue business as usual during the measurement period. They will receive the exact same intervention described above once data collection is complete.
  Interventions: Behavioral: Professional Development Enhancement

INTERVENTIONS:
Behavioral: Professional Development Enhancement — Professional development for SROs enhanced by content concerning trauma-informed care, cultural competency, restorative justice, and social-emotional learning.

SUMMARY:
The University of Florida's (UF) Lastinger Center for Learning, in partnership with the UF Psychology Department, have been funded by the National Institute of Justice to advance the skills of School Resource Officers (SROs) currently working in the Miami-Dade Schools Police Department through an innovative, scalable, online and in-person professional development system. The goal will be realized through a 36-month pilot project allowing for the development, testing, and refinement of the system conducted in partnership with the Miami-Dade County Public Schools, and includes an evaluation component to assess for efficacy and scalability.

DETAILED DESCRIPTION:
The University of Florida Lastinger Center for Learning and the Psychology Department aim to pilot-test a system of job-embedded professional development that will train Miami-Dade County SROs in research-based, best-practice techniques for addressing the unique needs of the school environment. Using a combination of both online and in-person supports this innovative approach to SRO professional development will provide programming that is highly impactful, easily accessible, and cost-effective to implement and eventually scale up nationally.

This goal will be realized through a 36-month pilot project allowing for the development, testing, and refinement of the system conducted in partnership with the Miami-Dade County Public Schools. Additionally, it includes an evaluation component to assess for efficacy and scalability.

Trainings will be comprised of online modules and expert coaching in the following four areas:

1. Social-Emotional Learning (SEL): to build student capacity using the Consortium of Academic & Social Emotional Learning's (CASEL) core competencies, including self- awareness, self-management, social awareness, responsible decision-making, and relationship skills; Many schools are implementing SEL program to manage disruptive behavior, reduce aggression, bullying, and other forms of school violence, and to promote positive interactions among all school members. SROs can play a critical role in reinforcing the skills taught in classrooms by modeling empathy, perspective-taking, positive coping strategies, adaptive problem-solving, emotional regulation, listening skills, problem-solving, and respectful behaviors when interacting with youth and other adults in the school building.
2. Trauma-Informed Care: to help officers understand and mitigate the neurological, biological, and psychological impact of trauma on affected children and adolescents' behavior; a trauma-informed approach acknowledges the centrality of trauma and its profound impact on students' perception of emotional and physical safety and relationships.
3. Cultural Competence/Implicit Bias/Intersectionality: to help SROs navigate the personal and structural racial and cultural barriers that students face as well as those specifically faced by lesbian, gay, bisexual, transgender, and questioning (LGBTQ) children and youth. More broadly, a lack of competence in working with LGBTQ and youth of color can lead to or exacerbate school violence and erode school climate.
4. Restorative Practices/Problem-Solving: to develop a school culture grounded in community problem-solving and productive restitution, as an alternative to punitive or retributive-based discipline. There are many practices that fall under the umbrella of Restorative Justice. Schools in the US have implemented a variety of restorative practices to address truancy, bullying, disciplinary issues, and interpersonal conflict. Restorative practices in schools can vary widely (i.e., conferencing, circles, mediation) but typically offer a dialogue between those who have harmed and those who have been harmed. The dialogue is intended to assist in working out restitution, holding individuals accountable, repairing the harm and their relationship, and reintegrating the person causing the harm back into the school community.

Procedure:

The research design for this project will be an experimental time-series design where 70 SROs are randomly assigned to participate in the program (Cohort 1), and a control group of 70 SROs is placed on a waiting list to participate in the program starting six months after the first group completes the program (Cohort 2). The design includes a short time-series with treatment and control SROs measured simultaneously at three waves. The three measurements will occur before treatment assignment, after the treatment group completes the program, and six months after participation. After these three measurements are taken, the control group will receive the program. According to sample size guidelines from CrimeSolutions.org, for a time-series design, a sample size of at least 51 is expected to allow detection of a medium effect (0.50). However, some SRO attrition from the program is expected, and the selected sample size of 70 per group will protect against excessive loss of power due to attrition. In this program, attrition will be minimized due to the individual work that each SRO will perform with a coach. Also, participants will receive multiple reminders of each content e-clinic, and participants that miss a live e-clinic will be contacted by their coaches to encourage viewing of the recorded version.

The assignment of SROs for the groups will be at the school level, where all SROs within a school will be placed in either the treatment or control groups. The rationale of a school-level assignment is to avoid spill-over effects between treated and control SROs in the same schools. The population of schools for this study will include middle and high schools, and the treatment and control groups will have SROs in middle and high schools at proportions similar to the population. Recruitment into the professional development and evaluation study will be coordinated among the project partners, the University of Florida and the Miami Dade Schools Police Department. Information will be sent out via email and presentations will be made at appropriate meetings to recruit potential participants.'

Professional Development Program Components:

1. E-Content Clinics- Content Clinics are offered online using digital video technology. The Clinics have two components - First, research-based content and practice relevant to the given subject or challenge; Second, actionable strategies for using this information to immediately improve instruction. The Clinics will be linked to coaching development with SRO sergeants so they can reinforce the lessons learned by their officers. Clinics will provide two-hour intensive opportunities for professional development four times a year. Each clinic will be offered online "live" and will also be recorded for later streaming to ensure maximum access. The Clinics will emphasize the current research on a topic as well as actionable strategies and techniques to use in schools. Clinics will also have short online quizzes to check learning.
2. Coaching- Coaching develops strong cadres of leaders that have profound expertise and substantial success in advancing teaching and learning outcomes. This approach uses existing personnel to reinforce and deepen learning through online professional development by embedding it in day-to-day activities. The UF Lastinger Center Coaching approach is built upon a set of foundational skills that will be applied to this project. In this model, SRO sergeants will be trained as coaches to help them bridge the content in the professional development sessions to the officers' daily work while also generally building their capacity to develop their direct reports. Coaching will provide: a) deeper understanding of the professional development content and how it will affect school safety; b) application of adult learning principles to support and enhance SRO practice; c) knowledge to plan and lead job-embedded professional development; d) the ability to use structured dialogue to support dynamic, fluid learning and strategy implementation to improve school safety. The energized pursuit of inquiry with SROs is to generate meaningful data to guide improvement. Upon completing the Coaching program, leaders/ supervisors of SROs will receive a certification from the Lastinger Center. They will also be able to schedule live video coaching sessions where they will work one-on-one with a Lastinger Center Master Coach to address a pressing issue, answer a question, or generally build the effectiveness of their practice. This will allow sergeants to participate in an evidence-based, collaborative coaching process and a supportive e-learning community regardless of their schedule.
3. Online Community of Practice- This scalable online platform allows users to create virtual communities of practice designed to strengthen the learning and collaboration network. A community of practice provides an online mentoring and professional development system to boost retention and accelerate the professional growth of SROs while simultaneously building the collaboration capacity and expertise of their coaches.

ELIGIBILITY:
Inclusion Criteria:

- Must be a School Resource Officer Employed by Miami-Dade County

Exclusion Criteria:

- Not being a School Resource Officer Employed by Miami-Dade County

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2019-08-09 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Change in knowledge of child development, classroom management, child problem behaviors, and behavior management strategies | Up to 52 weeks
  This assessment will be administered to all participant
  and non-participant SROs. The items will be developed by the study's team and evaluated using expert reviews and cognitive interviews. Following the first assessment, the discrimination of the items will be evaluated using item-to-total correlations and any items with low or negative item- to-total correlations will be removed from further use in the study.
Change in knowledge of Behavioral Principles as Applied To Children Test (KBPAC) - Short Form. | Up to 52 weeks
  The KBPAC is a 50-item instrument designed to measure basic knowledge of behavioral principles applied to children. The shortened 10-item version of the KBPAC had a Kuder-Richardson reliability estimate of 0.77 and was shown to have an internal reliability parallel to the 50-item, and 25-item versions of the test. Response options are correct or incorrect.
Change in Trauma-Informed Self-Assessment Test | Up to 52 weeks
  The TISAT was adapted from the Trauma- Informed Organizational Self-Assessment. The TISAT is a 17-item scale designed to measure an individual's knowledge of trauma-informed strategies associated with mental health outcomes, substance use, homelessness, triggers (reminders of traumatic events), and de-escalation techniques. Response options are a 6-point Likert-type scale where individuals self-report their level of confidence utilizing trauma-informed strategies.
Change in General Self-Efficacy Scale (GSE). | Up to 52 weeks
  The GSE is 10-item scale designed to measure self- reported self-efficacy. The instrument was found to be correlated with sentiments of positivity and work satisfaction with lower scores signaling stress, health complains, exhaustion, depression and anxiety. Response options range from "not at all true" to "exactly true."
Change in Self-Assessment of Social and Emotional Competencies (SASEC). | Up to 52 weeks
  The SASEC was adapted from Section 1-Part B of the "Self-Assessing Social and Emotional Instruction and Competencies: A tool for teachers". The measure is a self-report on a 4-point Likert-Type scale of how much individuals agree that they have specific social and emotional competencies influencing SRO's interactions at the school. The 21-item measure covers the following factors of Social Emotional Competencies: Self-Awareness, Self- Management/Emotion Regulation, Social Awareness, Relationship/Social Skills, and Responsible Decision Making.
Change in Intercultural Sensitivity Scale (ISS). | Up to 52 weeks
  The ISS is a 24-item measure of intercultural sensitivity through five factors: interaction engagement, respect of cultural differences, interaction confidence, interaction enjoyment, and interaction attentiveness. The self-reported instrument is measured in a 5-point Likert-Type scale (strongly disagree to strongly agree).
Change in Implicit Association Test (IAT). | Up to 52 weeks
  The Implicit Association Test measures implicit automatic associations by tracking the speed at which participants associate different groups of words. The scale is delivered electronically using an open-source software. Scores will be evaluated using the latest scoring procedure .
Change in LGBT Ally Identity Measure. | Up to 52 weeks
  The LGBT Ally Identity Measure is designed to evaluate the competencies of heterosexual allies of the LGBT community with four main factors: skills to support the LGBT community, awareness of LGBT oppression, knowledge of the LGBT experience, and engagement in action with LGBT members of the community. Response options range from "not at all true" to "very true for me." The 19-item scale had a Cronbach's alpha of .68 for the knowledge and skills subscale, .81 for the openness and support subscale, and .65 for the oppression awareness subscale .
Change in Measure of Role Clarity: | Up to 52 weeks
  Role clarity will be measured by five items, which have a five-point Liker scale from strongly disagree to strongly agree.
Change in Measure of Job Satisfaction | Up to 52 weeks
  The study team will measure general job satisfaction using a five-item short form of the Brayfield-Rothe job satisfaction scale. The items of this short form are: "Most days I am enthusiastic about my work," "I feel fairly satisfied with my present job," "I find real enjoyment in my work," "Each day at work seems like it will never end," and "I consider my job rather unpleasant." The last two items are reverse-scored.
Change in Measure of Intent to Quit | Up to 52 weeks
  The SROs intent to quit will be measure with two questions:
  1) How likely are you to quit your job within the next month? 2) How likely are you to quit your
  job within the next year? A five-point response scale will be used: "Very likely", "Somewhat likely", "Neither likely nor unlikely", "Somewhat unlikely", "Very unlikely".

CONTACTS AND LOCATIONS:
Overall Officials: Julia Graber, PhD, Principal Investigator — University of Florida
Locations (1):
- Miami Dade Public Schools, Miami, Florida, United States